CLINICAL TRIAL: NCT04820543
Title: Effects of Dose and Injection Site for Gummy Smile Treatment With Botulinum Type A: A Prospective Study
Brief Title: Effects of Dose and Injection Site for Gummy Smile Treatment With Botulinum Type A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Gong Xi, principal investigator, Peking University
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: pkussGS2
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Smiling; Botulinum Toxins, Type A
Keywords: gummy smile; botulinum toxin; dose and injection site
MeSH Terms: conditions — Smiling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and the outcomes assessor will be prevented from having knowledge of the interventions assigned to individual participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simplified Method (Experimental): In this method, a uniform BTX-A injection technique with single-site injection of 2 U BTX-A (total, 4 U) at both right and left levator labii superioris alaeque nasi muscles (LLSAN) was administered. The injection points located at the muscle bulge at the uppermost part of the nasolabial fold.
  Interventions: Drug: injection of Botulinum type A
- Individualized Method (Experimental): In this method, the patients were administered BTX-A after 8 months when the effect of the previous injection vanished. And A dosage and injection sites were individualized according to the degree of severity of anterior GE presented pretreatment. For mild GS (3 to< 5mm), 2 U BTX-A was injected at bilateral LLSAN. For moderate (5 to < 7mm) and severe GS (≥ 7mm), 3 U and 5 U of BTX-A were injected per side (total, 6 U and 10U). And The injection points located at both LLSAN and the Yonsei point, with half doses at each point.
  Interventions: Drug: injection of Botulinum type A

INTERVENTIONS:
Drug: injection of Botulinum type A — The participates were allocated to two different application methods: Simplified Method for the first injection and Individualized Method 8 months later. All the patients underwent twice injection with each methods with no change of the BTX-A(Botox, Allergan, Irvine, CA) and other injection details: Lyophilized 100 U of Botox was reconstituted in 2.5 mL of 0.9% sodium chloride solution. The injections were made with a 27-gauge insulin syringe. The treatment was an outpatient procedure and all injections were performed by one of the authors (X.G.). No anesthesia was given during the procedure.
  Other Names: injection of Botulinum type A(Botox, Allergan, Irvine, CA)

SUMMARY:
Botulinum type A (BTX-A) is an easy and efficacious treatment for gingival smile (GS). However, its dosage and injection sites effect among patients are controversial.The objective was to compare the reduction of gingival exposure using two methods in patients with different dosage and injection sites. In this prospective self-controlled study, healthy GS participates who had an anterior gingival exposure (GE) of more than 3 mm were enrolled and administered single-point injection of 2 U BTX-A per side in the Simplified Method. And after 8 months, the Individualized Method was administered with 2-5 U BTX-A (total, 4-10 U) injections into 1-2 points according to the severity presented pretreatment. Data were collected at baseline and 4, 12, and 32 weeks of follow-up.

DETAILED DESCRIPTION:
The smile is one of universal facial expressions of the humans. Gingival smile (GS) or gummy smile defined as any exposure of the gingiva >2 or 3 mm upon smiling, and can substantially vary from patient to patient, with patients presenting gummy exposures of up to more than 10 mm. The prevalence of GS is 10.57%, and it is more frequently seen in women. Although only an anatomical variation, it can be considered unattractive and cause significant distress and impact on one's quality of life. Moreover, most orthodontists and dentists regard GS as an important risk factors for dental treatment.

GS involves a complex interaction of facial muscles, bones and skin, specifically, it is related to the hypermobile upper lip (HUL) by the involved muscles and alterations in anatomical features such as short clinical dental crown, anterior dentoalveolar extrusion, maxillary excess and short upper lip. Therapies for GS range from botulinum toxin injections to surgical interventions according to its etiology. Whereas the outcomes of surgical procedures are long-lasting, botulinum toxin type A (BTX-A) treatment is an easy and fast outpatient procedure, requiring no downtime and with high efficacy rates. Nevertheless, there are controversies on the dosage and injection sites of BTX-A, and the efficiency of BTX-A for GS treatment shows great variation in different studies, with the improvement rate of gingival exposure (GE) ranging from 62.06% to 98%, Sucupira and Abramovitz advocate the use of an average amount of BTX-A of 2 U at bilateral levator labii superioris alaeque nasi muscles(LLSAN) for the treatment of GS, and an average satisfaction level of 9.75 on a 10-point scale was noted in their study. In their article, use of larger dosages and additional injection sites is discouraged: "Other target muscles described in the literature do not give any additional benefit to this application and could easily lead to lip ptosis, inferior lip protrusion, asymmetry, or excessive lengthening of the upper lip." Polo disagreed their argument. They believe that dosage and injection sites of BTX-A need to be individualized according to the degree of severity presented. However, no clinical study compared and verified their divergence, and the highly personal experience and uncertainty still limit the use of BTX-A for GS treatment. Some authors are of the opinion that injection with BTX-A is a safe and cosmetically effective treatment for GS only when performed by experienced practitioners. Other studies preferred to initiate the treatment with average-dose BTX-A injection to single sites initially, with retouching at a later stage, as and when required. Based on the lack of studies at the stage of creating the hypothesis for this study, the investigators compared the efficiency using the simplified method use of 2U BTX-A of at bilateral LLSAN and the individualized injection of dosage and injection sites according to the severity of anterior GS presented in patients, and also to assess safety and patients' satisfaction with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 3.0-mm anterior gingival exposure upon unrestricted, "full-blown" smiling
* healthy adults

Exclusion Criteria:

* contraindication of BTX-A
* previous diseases or treatments affecting the position of the gingiva or upper lips
* history of BTX-A injections to the head or neck region
* facial paralysis
* having received and/or receiving active orthodontic treatment that includes vertical dimension treatment, such as extrusion and intrusion, and presence of periodontal disease
* subject's refusal to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
anterior gingival exposure (GE) | 4 weeks postinjection
  The distance from the superior margin point of the right incisor to the lower margin of the upper lip upon maximum smile.

SECONDARY OUTCOMES:
bilateral posterior GE | 4 weeks postinjection
  The distance between the superior margin point of the right first premolars, the left first premolars and the lower margin of the upper lip, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University School and Hospital of Stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The investigators did not have the plan to make individual participant data available to other researchers.